CLINICAL TRIAL: NCT07061509
Title: Musculoskeletal and Cardiovascular Effects of Exercise Addiction in Recreational Bodybuilders
Brief Title: Exercise Addiction and Health Risks in Gym Users
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, ESRA PEHLIVAN, Principal Investigator, Saglik Bilimleri Universitesi
Other Study IDs: ExerciseAdd-1
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Exercise Addiction; Cardiovascular Abnormalities
MeSH Terms: conditions — Cardiovascular Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exercise-Dependent Group: Participants identified as "exercise dependent" based on scores from the Exercise Dependence Scale-21 (EDS-21). These individuals train at least 3 times per week and meet the criteria for exercise addiction.
  Interventions: Other: Battery of Physical and Psychological Assessments
- Non-Dependent Group: Participants who engage in regular resistance training (≥3 times/week) but do not meet the criteria for exercise addiction, based on EDS-21 scores.
  Interventions: Other: Battery of Physical and Psychological Assessments

INTERVENTIONS:
Other: Battery of Physical and Psychological Assessments — Participants in this observational study will not receive any therapeutic intervention. Instead, all individuals will undergo a series of standardized non-invasive assessments for data collection purposes. These include the Exercise Dependence Scale-21 (EDS-21) to classify exercise addiction status, the Drive for Muscularity Scale (DMS) to evaluate body image and muscle-related attitudes, and the Extended Nordic Musculoskeletal Questionnaire to determine the presence and severity of musculoskeletal symptoms. Cardiovascular risk will be assessed using the SCORE Risk Assessment System, which incorporates blood pressure, cholesterol, blood glucose, smoking status, and demographic data. Additional measurements will include oxygen saturation and heart rate using pulse oximetry, and blood pressure using a sphygmomanometer. These evaluations are intended solely for comparative analysis between exercise-dependent and non-dependent groups.

SUMMARY:
This observational study aims to investigate the prevalence of musculoskeletal injuries and cardiovascular risk factors among individuals with and without exercise addiction. Adult recreational gym users who have been engaging in resistance training for at least six months will be included. Participants will be divided into two groups based on their exercise dependence levels, and outcomes such as musculoskeletal symptoms, anabolic substance use, and cardiovascular risk scores will be compared between groups.

DETAILED DESCRIPTION:
The current study will examine the effects of exercise addiction on musculoskeletal and cardiovascular health in recreational gym users. Exercise addiction is characterized by compulsive training behavior despite physical or psychological harm and is increasingly prevalent among young adults, especially those engaged in bodybuilding.

Participants will be recruited from randomly selected fitness centers in Istanbul and categorized into exercise-dependent and non-dependent groups using the Exercise Dependence Scale-21 (EDS-21). Musculoskeletal symptoms will be assessed using the Extended Nordic Musculoskeletal Questionnaire. Cardiovascular risk will be evaluated using the SCORE Risk Assessment System, which considers factors such as blood pressure, smoking, cholesterol, and blood glucose levels. The Drive for Muscularity Scale (DMS) will also be applied to assess body image and muscle-related attitudes.

In addition to the physical assessments, participants will be asked about the use of anabolic steroids, and the frequency and patterns of such use will be recorded. The study will aim to raise awareness about the health consequences of excessive exercise and unregulated anabolic substance use, with the goal of informing preventive strategies and guiding future research.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Member of a fitness center
* Regular physical activity (≥3 times per week)
* Voluntary participation with informed consent

Exclusion Criteria:

* Diagnosed psychiatric illness
* Professional or elite athletes
* Incomplete questionnaire data

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of healthy adult individuals aged 18 years or older who are members of fitness centers in Istanbul and have been regularly engaging in resistance or bodybuilding training for at least six months. All participants must exercise at least three times per week and meet the inclusion criteria. Individuals will be divided into two groups based on their exercise dependence status: those who meet the criteria for exercise addiction and those who do not. Participants with professional athletic status or a diagnosed psychiatric illness will be excluded. The population represents recreational gym users with varying attitudes toward exercise behavior, body image, and supplement use, providing a real-world sample for assessing the musculoskeletal and cardiovascular impacts of exercise addiction.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Prevalence of musculoskeletal injuries | Baseline
  Assessment of musculoskeletal injuries and symptoms using the Extended Nordic Musculoskeletal Questionnaire.
Cardiovascular risk score | Baseline
  Evaluation of 10-year cardiovascular risk using the SCORE Risk Assessment System based on systolic blood pressure, smoking status, cholesterol, and blood glucose.

SECONDARY OUTCOMES:
Prevalence of anabolic steroid use | Baseline
  Self-reported use of anabolic agents, type, dose, and duration.
Exercise dependence level | Baseline
  Assessment via the Exercise Dependence Scale-21 (EDS-21).
Drive for muscularity | Baseline
  Assessment with the Drive for Muscularity Scale (DMS).

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Pehlivan, Istanbul, Üsküdar, Turkey (Türkiye)